CLINICAL TRIAL: NCT06082362
Title: Definition of a Personalized Signature of Chronic Inflammation and Early Aging Predictive of the Development of Comorbidities in Infertile Men
Brief Title: Personalized Signature of Chronic Inflammation and Early Aging Predictive of the Comorbidities in Infertile Men
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Salonia, Professor, IRCCS San Raffaele
Other Study IDs: PNRR-MAD-2022-12375994
Record Dates: First submitted 2023-06-13; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Male Infertility
Keywords: Infertility; Male Infertility; Comorbidity; Andrology; Immuno-epidemiology; Environmental factors; Genetic factors
MeSH Terms: conditions — Infertility, Male; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Infertile men: Men with infertility
  Interventions: Other: Collection of clinical and biological material
- Fertile men: Fertile men
  Interventions: Other: Collection of clinical and biological material
- Oncologic patients: Patients with kidney, bladder, chest, or pancreas tumors
  Interventions: Other: Collection of clinical and biological material

INTERVENTIONS:
Other: Collection of clinical and biological material — Collection of clinical and biological material (e.g., samples of semen, stool, urine, blood, buccal swab)

SUMMARY:
The aim of the project is identify new biomarkers and/or prognostic factors in order to develop personalized strategies to prevent the onset of tumor and/or non tumor comorbidity in infertile men.

DETAILED DESCRIPTION:
Infertility is a disease of nearly endemic proportions, affecting up to 15% of couples of reproductive ages. Overall, a pure male factor infertility underlies the problem in at least 30% of cases. General health status in infertile men is gaining increasing clinical attention throughout the last decades. Indeed, infertile men were shown to be at increased risk of nononcologic and oncologic morbidity and mortality compared to age-comparable fertile ones. Despite emerging and solid epidemiological studies, the common ground fostering overall health status and male infertility is still far from being understood. Notwithstanding the numerous hypotheses that have been considered to explain the potential link overall men's health status and male infertility - e.g., including genetic, endocrinological, and metabolic abnormalities - the exact nature of these associations remains unclear. Recent clinical findings showed evidence of onset of age-related comorbidities 10-15 years earlier in infertile compared to fertile men. Single-cell transcriptome profiling of testes of men with idiopathic germ cell aplasia revealed an immature testis with a somatic environment stuck at puberty with immaturity of Leydig cells associated with chronic tissue inflammation, fibrosis, and senescence phenotype of the somatic cells, as well markers of chronic inflammation in the blood. Compelling evidence indicate that defects in the regulatory arms of the immune system and metabolic status can be associated with the risk of developing numerous oncological and non-oncological diseases. Thus far, limited reliable data on the immunological status of infertile men are available. Preliminary data from the coordinating group of the project revealed increased pro-inflammatory cells and reduced T cells in peripheral blood of infertile men. Moreover, the few T cells observed in infertile men displayed an exhausted phenotype. The investigators proposed an innovative multidisciplinary approach to identify causal links between infertility as a disease and chronic inflammation and comorbidities. Moreover, the investigators aim at identifying novel prognostic biomarkers/tools toward the development of tailored prevention strategies of severe comorbidities in infertile men. They will combine extensive clinical data of a unique and homogenous cohort of infertile men and controls with state-of-the art transcriptomic approaches, a comprehensive monitoring and functional characterization of adaptive and innate immune cells, and the endocrine-metabolomic signature of men with primary infertility. The success of our strategy will be instrumental for defining novel molecular causes of male infertility, along with the pathophysiological mechanism behind the higher burden of comorbid conditions. Results will provide information on cell compartments, and the senescent and endocrine status, mostly in men with primary idiopathic infertility, and new insights into the etiology responsible for the early onset of comorbidities in infertile men. This will represent a breakthrough in the infertility field and a major advancement towards better caring of male patients and healthy ageing in the real-life setting and will set the stage for the development of more tailored clinical approaches to prevent malignant and nonmalignant comorbidities in infertile men. Thereof, the findings of the research project will have a significant rebound in terms of cost-effectiveness on the national health system.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 50 years;
* White race
* Men with OAT o iNOA infertility diagnosis
* ability to sign the consent information

Exclusion Criteria:

* inability to sign the consent information
* secondary infertility diagnosis
* history of hematological diseases
* people treated with antibiotics in the six months prior the enrollment

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertile men compared to fertile men and men with uro-oncologic tumors.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Endocrine-metabolomic parameters | Baseline
  Endocrine-metabolomic parameters from blood samples: Sex Hormone Binding Globulin (SHBG), 17 beta estradiol (E2), Follicle stimulating hormone (FSH), luteinizing hormone (LH), prolactin, thyroid-stimulating hormone (TSH), inhibin B, Anti-Muller Hormone (AMH), Glucose 6-phosphate Dehydrogenase (G6PD), parathyroid hormone (PTH), Vitamine D, blood glucose test, osteocalcin, Prostate Specific Antigen (PSA), albumin.
Functional characterization of immune cells | Baseline
  We will assess:
  * presence and frequency of different myeloid and lymphoid populations through a multi-color flow cytometry
  * the ability of Cluster of Differentiation CD4+ cells and of Cluster of Differentiation CD8+ T cells to proliferate and secrete cytokines in response to anti-Cluster of Differentiation CD3 monoclonal antibodies
  * the presence and concentration of cytokines and chemokines in the other leucocyte populations
  * Depth T cell compartments through a single cell RiboNucleic Acid-sequencing analysis
Clinical data | Baseline
  We will collect:
  * Clinical andrological and medical data through the physician's assessment
  * Body Mass Index (BMI)
  * waist circumference
  * a spermiogram analysis: the presence, the number, the motility, and the shape of spermatozoa

SECONDARY OUTCOMES:
Immunological outcomes | Baseline
  We will assess:
  * the activation of the inflammasome
  * IL-1ß/IL-18 release in response to Toll-like receptors stimulation through Enzyme-Linked Immunosorbent Assay
  * the expression of CASP1, NLRP3, AIM2, NLRC4, ASC, and IL1B genes through real-time PCR (polymerase chain reaction)
  We will assess:
  * the activation of the inflammasome
  * IL-1ß/IL-18 release in response to Toll-like receptors stimulation through Enzyme-Linked Immunosorbent Assay
  * the expression of CASP1, NLRP3, AIM2, NLRC4, ASC, and IL1B genes through real-time polymerase chain reaction (PCR)
Senescence biomarkers | Baseline
  We will assess:
  * senescence markers
  * mutations in a well-defined set of genes associated with normal ageing

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Salonia, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Lombardy, Italy